CLINICAL TRIAL: NCT05508399
Title: Predictive Biomarker Analysis and Model Construction of Tislelizumab Combined With Chemotherapy for Perioperative Treatment of G/GEJ Adenocarcinoma: A Single-center, Observational Study
Brief Title: Biomarker Analysis of Tislelizumab Combined With Chemotherapy for Perioperative Treatment of G/GEJ Adenocarcinoma
Status: Completed | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Gang Ji -2
Record Dates: First submitted 2022-08-17; First posted 2022-08-19 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-03

CONDITIONS: Locally Advanced Gastric Adenocarcinoma; PD-1
MeSH Terms: interventions — Sequence Analysis, RNA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biological samples of DNA will be collected before and after neoadjuvant treatment with PD-1 mab combined with chemotherapy, then they will be used to detect and analyze the variation in DNA. Biological samples of RNA detection will be used to analyze the expression profile. Combined with clinicopathological features, clinical treatment efficacy and prognosis, samples of DNA and RNA will be used to analyze biomarkers and construct models for predicting efficacy of PD-1 mab combined with chemotherapy in locally advanced gastric cancer. Meanwhile, the investigators are going to establish organoids with immune microenvironment from surgically resected tumor tissues of G/GEJ adenocarcinoma patients. Organoids will be treated with the same immune-chemotherapy drugs with the corresponding patients who accepted neoadjuvant therapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PD-1 group: Patients who are qualified for receiving anti-PD-1 antibody combined with chemotherapy neoadjuvant therapy
  Interventions: Other: DNA panel and RNA Sequencing

INTERVENTIONS:
Other: DNA panel and RNA Sequencing — Interventions include collecting samples, DNA panel test and full transcriptome sequencing.
  Before collecting samples, obtaining written informed consent from patient in advance.
  1. Blood cell samples;
  2. Paraffin sample of residual tumor tissue of biopsy;
  3. Paraffin sample of residual tumor tissue and paracancer tissue after gastrectomy.

SUMMARY:
G/GEJ adenocarcinoma is one of the most common malignant tumors in China, ranking the fifth highest incidence and third highest mortality worldwide. Currently, surgical resection is the preferred treatment for G/GEJ adenocarcinoma, while the 5-year survival rate of patients is lower than 25%. Compared with surgical resection, immunotherapy is proved to be able to effectively prolong the survival time of patients. On one hand, with the continuous promotion of immunotherapy drugs, the exploration of neoadjuvant application of immunotherapy in G/GEJ adenocarcinoma has become a hotspot in recent years. It's also on their way that clinical trials of programmed death receptor-1 (PD-1), programmed death ligand-1 (PD-L1) and other immune checkpoints are carried out. On the other hand, the research found that although the curative effect of immune therapy seems better, the present G/GEJ adenocarcinoma immunotherapy marker researches mainly focused on the late stage of the cancer, with few studies of immune markers of neoadjuvant therapy for G/GEJ adenocarcinoma. Additionally, it's not quite feasible for single biomarkers to predict the immune treatment effect precisely. Therefore, combined with clinicopathology and therapeutic effects, this study is aimed to construct the efficacy prediction model of anti-PD-1 antibody together with chemotherapy for G/GEJ adenocarcinoma, by detecting RNA expression. Furthermore, this study will perform drug sensitivity test and bio-molecular test on patient derived organoid model to validate the biomarkers found from biological specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80 (including 18 and 80);
2. G/GEJ adenocarcinoma confirmed by basic ultrasound gastroscopy, enhanced CT (PET/CT), MRI or diagnostic laparoscopy;
3. Biopsy histologically confirmed adenocarcinoma
4. As assessed by the investigator, patients who are qualified for receiving PD-1 mab combined with chemotherapy neoadjuvant therapy;
5. Patients who volunteer to participate in this study and sign the informed consent, with good compliance and cooperation in the acquisition of biological specimens.

Exclusion Criteria:

1. Patients whose biological specimens do not meet the detection standards;
2. In the judgment of the investigator, the patients with factors that might have caused the study to be terminated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with G/GEJ adenocarcinoma who are ready to receive PD-1 monoclonal antibody combined with chemotherapy neoadjuvant treatment.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-01-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Relative RNA biomarkers | From the initiation date of patients recruited into groups to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  At the RNA level, to identify the biomarkers related to the efficacy of neoadjuvant therapy with PD-1 mab combined with chemotherapy in locally advanced gastric cancer.
Prediction model for efficacy | From the date of completing collecting data, to the date of death from any cause or the end date of the whole trail, whichever came first, assessed up to 2 years
  A prediction model for the efficacy of PD-1 mab combined with chemotherapy, constructed on the basis of clinical pathology, gene variation, gene expression and other factors.

SECONDARY OUTCOMES:
Conditions of immune microenvironment | From the initiation date of patients recruited into groups to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  To monitor the changes of immune microenvironment before and after neoadjuvant treatment with PD-1 mab combined with chemotherapy for locally advanced gastric cancer. To evaluate whether the tumor infiltration immune cell and organoid co-cultural system can rebuild the tumor immune micro-environment, the immune cell subpopulations will be detected by single-cell sequencing, immunofluorescence staining and flow-cytometry.
Drug resistance mechanism | From the initiation date of patients recruited into groups to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  To explore the drug resistance mechanism of locally advanced gastric cancer after neoadjuvant therapy with PD-1 mab combined with chemotherapy.
Response of organoids to the same neoadjuvant drugs as the corresponding patients | From the initiation date of patients recruited into groups to the date of first documented progression or date of death from any cause, whichever came first, assessed up to 2 years
  The investigators will establish the G/GEJ adenocarcinoma organoid and tumor infiltration immune cell co-cultural model. The model will be treated with the same PD-1 mab combined with chemotherapy drugs as the corresponding patients. The viability of the organoids will be observed and quantified after treatment. The correlation of 3D organoid sensitivity and the patient response will be analyzed. And RNA expression detection of organoids before and after treatment will be performed to further validate the biomarkers from biological specimens.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi, China